CLINICAL TRIAL: NCT03958981
Title: The Use of Castor Oil for Induction of Labour in Women With Previous Caesarean Delivery: a Randomized Controlled Trial
Brief Title: Castror Oil for Labor Induction in Women With Previous Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Mohamed El Sharkawy (Unknown); Yomna Bayoumi (Unknown); mohamed hisham gouda (Unknown); Dina latif (Unknown)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: castor oil
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Induction of Labor
MeSH Terms: interventions — Castor Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- castor oil group (Experimental): 60 mL of castor oil in 140 mL of orange juice
  Interventions: Drug: Castor Oil
- placebo group (Placebo Comparator): Patients will receive sunflower oil as a placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Castor Oil — The intervention group will be given 60 mL of castor oil in 140 mL of orange juice
  Arms: castor oil group
Drug: placebo — the control group will be given a sunflower oil as a placebo with a similar texture to castor oil
  Arms: placebo group

SUMMARY:
Nowadays, more and more women embark on pregnancy with previous Caesarean scar. One in five pregnancies requires induction of labour. The use of non-pharmacological methods (methods without using medication) has been gaining popularity for women who are not good candidates, such as women with previous Caesarean scar, for induction with medications such as prostaglandin. Labour induction with prostaglandin carries a higher risk of uterine rupture and thus it is not routinely offered to women with previous Caesarean delivery in Cairo University Hospital. Non-pharmacological methods of induction of labour appear to be safe in women with previous Caesarean delivery. However, various methods are available and the efficacy among them remain in doubt.

DETAILED DESCRIPTION:
In Cairo University Hospital, castor oil, which is a type of induction methods, is routinely offered to women with previous Caesarean delivery who require induction of labor. However, castor oil may not exert its labor induction effect immediately and the delivery may be delayed by up to 8 days. This may render a proportion of women resort to repeated Caesarean section for failed induction. Castor oil is traditionally given by midwives in order to induce labor.

The investigators are intent to recruit 70 healthy pregnant women with a history of previous one cesarean section and with no contraindication to trial of labor after cesarean . Women will be randomly and blindly divided into equal-sized intervention group and control group. Intervention group will be given a single dose 60 mL of castor oil in 140 mL of orange juice, while control group will be given a placebo with similar texture. Primary outcomes to be tested are the percentage of women entering active labor within 24 hours of castor oil or placebo administration and the number of successful vaginal deliveries after cesarean.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with one previous lower segment Caesarean section who are admitted to Cairo University Hospital for induction of labor (IOL) will be recruited. The inclusion criteria are age at least 20 years old, gestational age at recruitment from 36 weeks to 38 weeks ±6 days, gestational age at induction= 39 weeks, singleton pregnancy, reassuring fetal status, and Bishop score ≤ 6.

Exclusion Criteria:

* Prior high-risk uterine scar; uterine rupture, classical CS, hysterotomy, or myomectomy
* Short inter-delivery interval (<12 months)
* Complications in the previous CS (e.g. puerperal sepsis)

Obstetric indication for CS (either elective or emergency):

* Placenta praevia
* Placental abruption
* Documented evidence of cephalopelvic disproportion
* Fetal macrosomia (estimated fetal weight >4 kg)
* Fetal anomalies interfering with vaginal delivery e.g. hydrocephalus
* Fetal distress or non-reassuring Cardiotocography pattern

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Percentage of women entering active phase within 24 hours of administering castor oil/placebo | two weeks
  Actual time of delivery
number of successful VBAC cases | 24 hours
  number of successful cases who delivered vaginally

SECONDARY OUTCOMES:
Neonatal apgar scores | 1 minute and 5 minute after delivery
  Neonatal APGAR scores
Neonatal complications including hospitalization in NICU | immediately after birth
  Were there any admissions to NICU, what was the reason ?
Mode of delivery (ie. Normal delivery Vs. Cesarean delivery) | Within two weeks of enrollment
  Mode of delivery
duration of labor | 24 hours
  duration of labor in hours
number of cases needing oxytocin augmentation | 24 hours
  number of cases needing oxytocin augmentation

CONTACTS AND LOCATIONS:
Overall Officials: Yomna Bayoumi, MD, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine Cairo university, Cairo, Egypt